CLINICAL TRIAL: NCT05358275
Title: The Evaluation of the Effect of Performing Guided Lid Surgery With Enucleation of Cystic Lesions Compared to Conventional Cystic Enucleation; a Randomized Clinical Trial
Brief Title: The Evaluation of the Effect of Performing Guided Lid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28-4-2022 OMFS
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Odontogenic Cysts
MeSH Terms: conditions — Odontogenic Cysts

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 1:1 allocation ratio
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Guided lid surgery is performed to reduce the loss of bone post operative
  Interventions: Device: surgical cutting guide with piezo
- control group (Active Comparator): The patient will receive active ordinary treatment for removal of odontogenic cysts
  Interventions: Other: control

INTERVENTIONS:
Device: surgical cutting guide with piezo — 3D planned lid surgery
  Arms: study group
Other: control — ordinary cyst enucleation
  Arms: control group

SUMMARY:
to evaluate the percentage of bone volume regain along with postoperative pain in cases done using the bone lid technique in comparison with those done using the conventional cyst enucleation technique.

DETAILED DESCRIPTION:
The study will involve eighteen patients selected from the outpatient clinic, Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Ain Shams University.

The patients included in this study will be informed about the full details of this research and they will sign an informed consent. Moreover, this research will be reviewed by the research ethics committee, Faculty of Dentistry, Ain Shams University.

Randomization:

The study consists of two groups each containing 10 patients. Patients will be randomly allocated according to predetermined computer-generated randomization using (www.randomizer.org).

PICO:

P: Patients with expansile cystic lesions with intact bony cortex of a minimum 1mm thickness.

I: Cyst enucleation using the bone lid technique and piezoelectric device. C: Cyst enucleation using the conventional buccal bone ostectomy technique. O: Percentage of bone volume recovery. T: 6 months postoperative.

Inclusion criteria:

1. Age ranging from 18-60 years.
2. Have free medical history or controlled systemic disease.
3. Expansile cystic lesion with intact cortical bone extending from 2-6 teeth.
4. A minimum thickness of 1 mm of the cortical bone.

Exclusion criteria:

1. Patients with history of surgery in the area affected by the cystic lesion.
2. Patients with suspected malignant tumors in the area.

Pre-operative assessment:

Proper history is obtained followed by palpation of the affected area to check tenderness or suspected superimposed infection. Aspiration biopsy is done to ensure the nature of the lesion being cystic. Cone Beam Computed Tomography (CBCT) is done to assess the exact size of the lesion and plan for the surgical cutting guide.

Patients with intact cortical bone related to the cystic lesion will be enrolled in this study. All patients will receive full information about the procedures where the risks and benefits will be thoroughly explained to them. They will then be asked to give their consent.

Sample size calculation:

Considering that there was around 93% difference between the cystic cavity before and after lid surgery with enucleation (19). After setting the α at 0.05 and β at 0.2; the minimal sample size was calculated and revealed that the minimum number to achieve statistical data was 10 patients in each goup (total number of patients= 20).

Pre-operative patient preparation:

1. Fasting for 6-8 hours before the procedure.
2. Laboratory investigations to assess his/ her medical condition if the procedure is to be performed under general anesthesia;

   * Complete blood count (CBC).
   * Bleeding profile; PT, PTT, INR.
   * Liver function test.
   * Kidney function test.
   * Blood sugar level; fasting and 2-hours post-brandial.

Surgical procedure:

Anesthetizing the surgical area is done using the selected suitable nerve block technique with articaine 4% and 1:100,000 epinephrine.

1. Flap reflection:

   A full thickness muco-periosteal flap is reflected using no.15 blade. The extent of the flap incisions shall involve one tooth mesial to the lesion and one tooth distal to the lesion.
2. Surgical guide fixation:

   The surgical cutting guide is adapted in place and fixed using micro-screws to ensure proper stability of the guide and accuracy of the bony window.
3. Bone lid fabrication:

   The bony window is cut guided by the edges in the cutting guide using piezoelectric device under copious irrigation. The window is then dissected bluntly from the attached cystic lesion using a muco-periosteal elevator and a bone curette.
4. Enucleation of the cystic lesion:

   The lesion is carefully separated from the surrounding bone using a muco-periosteal elevator and a bone curette while being held with a toothed tissue forceps or Allis forceps. The excised lesion will be placed in a jar containing 10% formaldehyde to be sent to the Oral Pathology lab for excisional biopsy confirmation of the nature of the lesion. This is followed by careful curettage of the surgical bed to ensure absence of any remnants of the lesion followed by rinsing using isotonic saline solution.
5. Fixation of the bone lid:

   The previously removed bone lid is reoriented back in place and fixed using 2.3 micro-plates and micro-screws for rigid fixation.
6. Closure of the flap:

The flap is sutured using 4-0 vicryl resorbable suture to achieve primary closure.

The control group will be done using the conventional buccal ostectomy technique by reflection of a full thickness mucoperiosteal flap followed by removal of part of the cortical bone to allow enough access to the cystic lesion. The lesion is enucleated afterwards by removing the entire lining and the flap is closed at the end of the procedure using 4-0 vicryl resorbable suture. No surgical guide is used and the removed part of the cortical bone is grinded using a high speed handpiece, a rounded surgical bur and a bone curette.

Immediate post-operative medications:

1. Amoxicillin/ clavulanate 1gm tablets every 12 hours for 5 days.
2. Chymotrypsin 300E.A.U. 2 tablets every 8 hours for 5 days.
3. Ibuprofen 600mg tablets every 12 hours for 5 days.

Immediate post-operative instructions:

1. Avoid vigorous rinsing or spitting for the first 24 hours.
2. Place ice packs over the surgical area for 10 minutes and repeated every 30 minutes over the first 6 hours.
3. Avoid hot, hard or crunchy food for the first 3 days.
4. After 24 hours, start rinsing with warm isotonic saline solution 3 times per day for 7 days.
5. After 24 hours, start placing warm packs over the surgical area 3 times per day for 7 days.

Follow up:

1. Percentage of bone volume regained will be evaluated using CBCT 6 months after the intervention (a total of 2 CBCTs; one pre-operative and one 6 months post-operative).
2. Pain will be assessed immediately postoperative and after 6 months by Visual Analog Scale from (0-10), as 0 means absence of pain and 10 means maximum pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18-60 years.
2. Have free medical history or controlled systemic disease.
3. Expansile cystic lesion with intact cortical bone extending from 2-6 teeth.
4. A minimum thickness of 1 mm of the cortical bone.

Exclusion Criteria:

1. Patients with history of surgery in the area affected by the cystic lesion.
2. Patients with suspected malignant tumors in the area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Regain of bone volume | 6 months
  evaluation of formed bone using CBCT

SECONDARY OUTCOMES:
Pain with visual analogue scale | one week
  evaluation of pain by exposing patient to a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: mohamed diaa, Study Chair — Ain Shams University
Locations (1):
- Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No